CLINICAL TRIAL: NCT02102932
Title: Relative Bioavailability of Empagliflozin (12.5 or 5 mg)/Metformin (850 mg or 500 mg) Fixed Dose Combination Tablets Compared to Single Tablets Administered Together to Healthy Chinese Male and Female Volunteers in an Open-label, Randomised, Single-dose, Two-way Crossover Study
Brief Title: Bioavailability of Empagliflozin/Metformin Fixed Dose Combinations (FDCs) in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1276.23
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Metformin

ARMS (4):
- 12.5 mg empagliflozin/850 mg metformin (Experimental): 24 subjects (12 male and 12 female) will be assigned to 2 treatment sequences. cross-over design was adopted to ensure each patient would take fixed dose combination tablets of 12.5 mg empagliflozin/850 mg metformin and single 10 mg empagliflozin, 2.5 mg empagliflozin, 850 mg metformin tablets single dose in randomized order
  Interventions: Drug: 12.5 mg empagliflozin; Drug: 850 mg metformin; Drug: 12.5 mg empagliflozin/850 mg metformin FDC
- 5 mg empagliflozin/850 mg metformin (Experimental): 24 subjects (12 male and 12 female) will be assigned to 2 treatment sequences. cross-over design was adopted to ensure each patient would take fixed dose combination tablets of 5 mg empagliflozin/850 mg metformin and single Empagliflozin(5mg) and metformin (850mg) tablets single dose in randomized order
  Interventions: Drug: 5 mg empagliflozin/850 mg metformin FDC; Drug: 5 mg empagliflozin; Drug: 850 mg metformin
- 12.5 mg empagliflozin/500 mg metformin (Experimental): 24 subjects (12 male and 12 female) will be assigned to 2 treatment sequences. cross-over design was adopted to ensure each patient would take fixed dose combination tablets of 12.5 mg empagliflozin/500 mg metformin and single 10 mg empagliflozin, 2.5 mg empagliflozin, 500 mg metformin tablets single dose in randomized order
  Interventions: Drug: 12.5 mg empagliflozin; Drug: 12.5 mg empagliflozin/500 mg metformin FDC; Drug: 500 mg metformin
- 5 mg empagliflozin/500 mg metformin (Experimental): 24 subjects (12 male and 12 female) will be assigned to 2 treatment sequences. cross-over design was adopted to ensure each patient would take fixed dose combination tablets of 5 mg empagliflozin/500 mg metformin and single Empagliflozin(5mg) and metformin (500mg) tablets single dose in randomized order
  Interventions: Drug: 5 mg empagliflozin; Drug: 5 mg empagliflozin/500 mg metformin FDC; Drug: 500 mg metformin

INTERVENTIONS:
Drug: 5 mg empagliflozin/850 mg metformin FDC — 5 mg empagliflozin/850 mg metformin FDC
  Arms: 5 mg empagliflozin/850 mg metformin
Drug: 12.5 mg empagliflozin — 10 mg empagliflozin tablet and 2.5 mg empagliflozin tablet
  Arms: 12.5 mg empagliflozin/500 mg metformin
Drug: 12.5 mg empagliflozin — 10mg empagliflozin tablet and 2.5 mg empagliflozin tablet
  Arms: 12.5 mg empagliflozin/850 mg metformin
Drug: 850 mg metformin — 850mg metformin tablet
  Arms: 12.5 mg empagliflozin/850 mg metformin
Drug: 5 mg empagliflozin — 5 mg empagliflozin
  Arms: 5 mg empagliflozin/850 mg metformin
Drug: 5 mg empagliflozin — 5 mg empagliflozin
  Arms: 5 mg empagliflozin/500 mg metformin
Drug: 850 mg metformin — 850 mg metformin
  Arms: 5 mg empagliflozin/850 mg metformin
Drug: 12.5 mg empagliflozin/850 mg metformin FDC — 12.5 mg empagliflozin/850 mg metformin FDC
  Arms: 12.5 mg empagliflozin/850 mg metformin
Drug: 12.5 mg empagliflozin/500 mg metformin FDC — 12.5 mg empagliflozin/500 mg metformin FDC
  Arms: 12.5 mg empagliflozin/500 mg metformin
Drug: 5 mg empagliflozin/500 mg metformin FDC — 5 mg empagliflozin/500 mg metformin FDC
  Arms: 5 mg empagliflozin/500 mg metformin
Drug: 500 mg metformin — 500 mg metformin
  Arms: 12.5 mg empagliflozin/500 mg metformin
Drug: 500 mg metformin — 500 mg metformin
  Arms: 5 mg empagliflozin/500 mg metformin

SUMMARY:
The aim of the trial is to assess the relative bioavailability of fixed dose combination tablets of Empagliflozin and metformin compared to the administration of single tablets (Empagliflozin and metformin ) in Chinese subjects. The availability of a fixed dose combination tablet is expected to significantly enhance patient's compliance with antidiabetic treatment, in particular with concern to the frequent polypharmacy in diabetic patients.

ELIGIBILITY:
Inclusion criteria:

Healthy male and female subjects

Exclusion criteria:

Any relevant deviation from healthy conditions

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1276.23.86002 Boehringer Ingelheim Investigational Site, Beijing, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed as an open-label, randomised, single-dose, two-way crossover trial consisting of four trial parts. In each trial part the aim was to investigate the relative bioavailability of the Test treatment (T) and to compare it with the Reference treatment (R).
Groups:
- T1R1: Study Part 1:
  T1: Oral administration of a single fixed dose combination (FDC) tablet 12.5 mg empagliflozin/850 mg metformin R1: Oral administration of 1 tablet empagliflozin 10 mg + 1 tablet empagliflozin 2.5 mg + 1 tablet Glucophage® 850 mg; A washout period of at least 7 days was to be maintained between T1 and R1.
- R1T1: Study Part 1:
  R1: Oral administration of 1 tablet empagliflozin 10 mg + 1 tablet empagliflozin 2.5 mg + 1 tablet Glucophage® 850 mg T1: Oral administration of a single FDC tablet 12.5 mg empagliflozin/850 mg metformin; A washout period of at least 7 days was to be maintained between R1 and T1.
- T2R2: Study Part 2:
  T2: Oral administration of a single FDC tablet 5 mg empagliflozin/850 mg metformin R2: Oral administration of 1 tablet empagliflozin 5 mg + 1 tablet Glucophage® 850 mg; A washout period of at least 7 days was to be maintained between T2 and R2.
- R2T2: Study part 2:
  R2: Oral administration of 1 tablet empagliflozin 5 mg + 1 tablet Glucophage® 850 mg; T2: Oral administration of a single FDC tablet 5 mg empagliflozin/850 mg metformin; A washout period of at least 7 days was to be maintained between R2 and T2.
- T3R3: Study Part 3:
  T3: Oral administration of a single FDC tablet 12.5 mg empagliflozin/500 mg metformin R3: Oral administration of 1 tablet empagliflozin 10 mg + 1 tablet empagliflozin 2.5 mg + 1 tablet Glucophage® 500 mg; A washout period of at least 7 days was to be maintained between T3 and R3.
- R3T3: Study Part 3:
  R3: Oral administration of 1 tablet empagliflozin 10 mg + 1 tablet empagliflozin 2.5 mg + 1 tablet Glucophage® 500 mg T3: Oral administration of a single FDC tablet 12.5 mg empagliflozin/500 mg metformin; A washout period of at least 7 days was to be maintained between R3 and T3
- T4R4: Study Part 4:
  T4: Oral administration of a single FDC tablet 5 mg empagliflozin/500 mg metformin R4: Oral administration of 1 tablet empagliflozin 5 mg + 1 tablet Glucophage® 500 mg; A washout period of at least 7 days was to be maintained between T4 and R4.
- R4T4: Study Part 4:
  R4: Oral administration of 1 tablet empagliflozin 5 mg + 1 tablet Glucophage® 500 mg; T4: Oral administration of a single FDC tablet 5 mg empagliflozin/500 mg metformin; A washout period of at least 7 days was to be maintained between R4 and T4
Period: Overall Study
Arm/Group | T1R1 | R1T1 | T2R2 | R2T2 | T3R3 | R3T3 | T4R4 | R4T4
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who were dispensed study medication and were documented to have received at least 1 dose of trial medication
Groups:
- Total: Total of all reporting groups
Arm/Group | T1R1 | R1T1 | T2R2 | R2T2 | T3R3 | R3T3 | T4R4 | R4T4 | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (4.8) | 27.0 (5.3) | 26.8 (5.3) | 24.3 (3.4) | 24.8 (4.3) | 24.4 (3.9) | 24.6 (3.7) | 25.6 (4.8) | 25.5 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 7 | 5 | 5 | 7 | 5 | 7 | 48
  Male | 5 | 7 | 5 | 7 | 7 | 5 | 7 | 5 | 48

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-∞) for Empagliflozin
Description: Area under the concentration-time curve of the empagliflozin in plasma over the time interval from 0 extrapolated to infinity
Time Frame: 1 hour (h) before drug administration and 20 min (m), 40m, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after drug administration
Population: Pharmacokinetic set (PKS):
  The PKS included all evaluable subjects of the TS who provided at least 1 observation for at least 1 primary PK endpoint in both treatment periods without Important protocol violations (IPV) relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol * h/L
Groups:
- T1 (FDC): Oral administration of a single fixed dose combination (FDC) tablet 12.5 mg empagliflozin/850 mg metformin
- R1 (FC): Oral administration of free combination (FC) of 1 tablet empagliflozin 10 mg + 1 tablet empagliflozin 2.5 mg + 1 tablet Glucophage® 850 mg
- T2 (FDC): Oral administration of a single FDC tablet 5 mg empagliflozin/850 mg metformin
- R2 (FC): Oral administration of FC of 1 tablet empagliflozin 5 mg + 1 tablet Glucophage® 850 mg
- T3 (FDC): Oral administration of a single FDC tablet 12.5 mg empagliflozin/500 mg metformin
- R3 (FC): Oral administration of FC of 1 tablet empagliflozin 10 mg + 1 tablet empagliflozin 2.5 mg + 1 tablet Glucophage® 500 mg
- T4 (FDC): Oral administration of a single FDC tablet 5 mg empagliflozin/500 mg metformin
- R4 (FC): Oral administration of FC of 1 tablet empagliflozin 5 mg + 1 tablet Glucophage® 500 mg
Arm/Group | T1 (FDC) | R1 (FC) | T2 (FDC) | R2 (FC) | T3 (FDC) | R3 (FC) | T4 (FDC) | R4 (FC)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
nmol * h/L | 4330 (16.6) | 4110 (15.3) | 1680 (22.0) | 1630 (21.1) | 4200 (20.3) | 4060 (18.6) | 1610 (16.5) | 1560 (17.7)
Statistical Analysis 1: Comparison: T1 (FDC) vs R1 (FC); The statistical model used was an analysis of variance (ANOVA) model on the logarithmic scale. This model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 105.29, 90% CI 2-sided [101.92 to 108.78], Standard Deviation 6.6 — Ratio of the geometric means for treatments (Test (T1) versus Reference (R1)) i.e. T1/R1. The standard deviation is actually the intra-individual gCV
Statistical Analysis 2: Comparison: T2 (FDC) vs R2 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 103.23, 90% CI 2-sided [99.91 to 106.65], Standard Deviation 6.6 — Ratio of the geometric means for treatments (Test (T2) versus Reference (R2)) i.e. T2/R2. The standard deviation is actually the intra-individual gCV
Statistical Analysis 3: Comparison: T3 (FDC) vs R3 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 103.56, 90% CI 2-sided [99.73 to 107.54], Standard Deviation 7.6 — Ratio of the geometric means for treatments (Test (T3) versus Reference (R3)) i.e. T3/R3. The standard deviation is actually the intra-individual gCV
Statistical Analysis 4: Comparison: T4 (FDC) vs R4 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 102.81, 90% CI 2-sided [99.36 to 106.37], Standard Deviation 6.9 — Ratio of the geometric means for treatments (Test (T4) versus Reference (R4)) i.e. T4/R4. The standard deviation is actually the intra-individual gCV

2. Primary Outcome: AUC(0-∞) for Metformin
Description: Area under the concentration-time curve of the metformin in plasma over the time interval from 0 extrapolated to infinity
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng * h/mL
Arm/Group | T1 (FDC) | R1 (FC) | T2 (FDC) | R2 (FC) | T3 (FDC) | R3 (FC) | T4 (FDC) | R4 (FC)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
ng * h/mL | 11600 (18.9) | 11100 (17.4) | 11700 (21.8) | 11000 (24.0) | 7800 (18.9) | 7510 (17.8) | 7030 (20.7) | 7340 (18.8)
Statistical Analysis 1: Comparison: T1 (FDC) vs R1 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 104.56, 90% CI 2-sided [97.56 to 112.07], Standard Deviation 14.0 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: T2 (FDC) vs R2 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 105.80, 90% CI 2-sided [99.32 to 112.70], Standard Deviation 12.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: T3 (FDC) vs R3 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 103.75, 90% CI 2-sided [98.18 to 109.63], Standard Deviation 11.2 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: T4 (FDC) vs R4 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 95.77, 90% CI 2-sided [89.88 to 102.03], Standard Deviation 12.8 — [estimate comment as in outcome 1, analysis 4]

3. Primary Outcome: Cmax for Empagliflozin
Description: Maximum measured concentration of the empagliflozin in plasma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | T1 (FDC) | R1 (FC) | T2 (FDC) | R2 (FC) | T3 (FDC) | R3 (FC) | T4 (FDC) | R4 (FC)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
nmol/L | 644 (18.2) | 605 (15.3) | 263 (17.7) | 237 (20.7) | 569 (22.1) | 561 (25.3) | 228 (16.4) | 221 (22.2)
Statistical Analysis 1: Comparison: T1 (FDC) vs R1 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 106.44, 90% CI 2-sided [100.44 to 112.80], Standard Deviation 11.8 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: T2 (FDC) vs R2 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0021, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 110.78, 90% CI 2-sided [103.80 to 118.24], Standard Deviation 13.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: T3 (FDC) vs R3 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 101.38, 90% CI 2-sided [94.82 to 108.39], Standard Deviation 13.6 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: T4 (FDC) vs R4 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 103.02, 90% CI 2-sided [95.08 to 111.63], Standard Deviation 16.3 — [estimate comment as in outcome 1, analysis 4]

4. Primary Outcome: Cmax for Metformin
Description: Maximum measured concentration of the metformin in plasma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | T1 (FDC) | R1 (FC) | T2 (FDC) | R2 (FC) | T3 (FDC) | R3 (FC) | T4 (FDC) | R4 (FC)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
ng/mL | 1920 (20.9) | 1830 (16.6) | 1950 (26.4) | 1840 (26.0) | 1290 (22.2) | 1230 (27.1) | 1150 (25.5) | 1190 (21.3)
Statistical Analysis 1: Comparison: T1 (FDC) vs R1 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 104.91, 90% CI 2-sided [99.29 to 110.86], Standard Deviation 11.2 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: T2 (FDC) vs R2 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0008, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 106.32, 90% CI 2-sided [98.39 to 114.88], Standard Deviation 15.7 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: T3 (FDC) vs R3 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0003, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 104.44, 90% CI 2-sided [96.68 to 112.82], Standard Deviation 15.7 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: T4 (FDC) vs R4 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0004, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 96.61, 90% CI 2-sided [88.90 to 104.99], Standard Deviation 16.9 — [estimate comment as in outcome 1, analysis 4]

5. Secondary Outcome: AUC(0-tz) of Empagliflozin
Description: Area under the concentration-time curve of the empagliflozin in plasma over the time interval from 0 up to the last quantifiable data point
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol * h/L
Arm/Group | T1 (FDC) | R1 (FC) | T2 (FDC) | R2 (FC) | T3 (FDC) | R3 (FC) | T4 (FDC) | R4 (FC)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
nmol * h/L | 4270 (16.6) | 4060 (14.7) | 1650 (21.5) | 1600 (21.0) | 4140 (19.7) | 4010 (18.5) | 1580 (16.7) | 1540 (17.7)
Statistical Analysis 1: Comparison: T1 (FDC) vs R1 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 105.16, 90% CI 2-sided [101.97 to 108.45], Standard Deviation 6.2 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: T2 (FDC) vs R2 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 103.07, 90% CI 2-sided [99.75 to 106.50], Standard Deviation 6.6 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: T3 (FDC) vs R3 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 103.14, 90% CI 2-sided [99.37 to 107.04], Standard Deviation 7.5 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: T4 (FDC) vs R4 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 102.61, 90% CI 2-sided [99.10 to 106.25], Standard Deviation 7.0 — [estimate comment as in outcome 1, analysis 4]

6. Secondary Outcome: AUC(0-tz) of Metformin
Description: Area under the concentration-time curve of the metformin in plasma over the time interval from 0 up to the last quantifiable data point
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng* h/mL
Arm/Group | T1 (FDC) | R1 (FC) | T2 (FDC) | R2 (FC) | T3 (FDC) | R3 (FC) | T4 (FDC) | R4 (FC)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
ng* h/mL | 11400 (19.2) | 10800 (17.6) | 11400 (23.1) | 10800 (25.1) | 7630 (18.9) | 7420 (17.9) | 6790 (24.7) | 7230 (18.3)
Statistical Analysis 1: Comparison: T1 (FDC) vs R1 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 105.33, 90% CI 2-sided [99.34 to 111.68], Standard Deviation 11.9 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: T2 (FDC) vs R2 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 105.75, 90% CI 2-sided [99.09 to 112.85], Standard Deviation 13.2 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: T3 (FDC) vs R3 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 102.90, 90% CI 2-sided [97.11 to 109.03], Standard Deviation 11.7 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: T4 (FDC) vs R4 (FC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANOVA — P-value for ratio outside interval 80-125; Ratio of the geometric means = 93.84, 90% CI 2-sided [87.74 to 100.36], Standard Deviation 13.6 — [estimate comment as in outcome 1, analysis 4]

ADVERSE EVENTS:
Time Frame: First drug administration until 7 days after last drug administration, up to 8 days
Arm/Group | T1 (FDC) | R1 (FC) | T2 (FDC) | R2 (FC) | T3 (FDC) | R3 (FC) | T4 (FDC) | R4 (FC)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 8/24 | 8/24 | 9/24 | 11/24 | 12/24 | 11/24 | 7/24 | 9/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T1 (FDC) (N=24) | R1 (FC) (N=24) | T2 (FDC) (N=24) | R2 (FC) (N=24) | T3 (FDC) (N=24) | R3 (FC) (N=24) | T4 (FDC) (N=24) | R4 (FC) (N=24)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1 | 2 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 7 | 11 | 10 | 8 | 3 | 5
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 1 | 1 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 3
Blood bilirubin unconjugated increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Glucose urine present (Investigations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights